CLINICAL TRIAL: NCT06734390
Title: Management of Patients Under 18 Years of Age Who Have Had Bladder Neck Procedures
Brief Title: Bladder Neck Surgery in Children with Neurogenic Bladder
Acronym: CERPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, Destinval Christelle, M.D., University Hospital, Clermont-Ferrand
Other Study IDs: M24DC1103
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Incontinence; Bladder Dysfunction; Spina Bifida; Neurogenic Bladder Disorder; Child, Only
Keywords: Bladder Neck Surgery; Surgical Outcomes; Child; Retrospective Study
MeSH Terms: conditions — Spinal Dysraphism; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Bladder Neck Surgery — Bladder Neck Surgery regroups many surgical procedures to cure urinary incontinence.

SUMMARY:
Surgical outcomes of bladder neck surgery in children with neurogenic bladder. Consequences on bladder voiding.

DETAILED DESCRIPTION:
Surgical outcomes of bladder neck surgery in children with neurogenic bladder:

Quality of voiding: spontaneous, need for catheterization, or incontinence. Other surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurogenic bladder and younger than 18 years old , who underwent a bladder neck procedure

Exclusion Criteria:

* Patients, with neurogenic bladder and older than 18 years old ,who underwent a bladder neck procedure

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with neurogenic bladder
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with delayed or incomplete opening of the bladder neck during the voiding phase of micturition impeding urine flow | Before surgery
  Abdominal ultrasound, cysto-urethrogram and uroflowmetry help diagnose delayed or incomplete opening of the bladder neck.
Long-term urinary continence | Through study completion, an average of 2 years
  Reporting if the patients are dry or need catheterizations or protections

SECONDARY OUTCOMES:
Length of stay | From admission to discharge home, up to 20 days
  Length of stay
Complications after bladder neck procedure | Through study completion, an average of 2 years
  bleeding, bowel obstruction, surgical hernia, urinary stone, urinary infection
Follow-up | Through study completion, an average of 2 years
  The time length between the surgery date and the postoperative consultation date.
  Follow-up represents the time between the surgery and postoperative consultation dates in days, months, or years.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization, the investigators won't share individual participant data

REFERENCES:
- [Background] Stein R, Bogaert G, Dogan HS, Hoen L, Kocvara R, Nijman RJM, Quaedackers J, Rawashdeh YF, Silay MS, Tekgul S, Radmayr C. EAU/ESPU guidelines on the management of neurogenic bladder in children and adolescent part II operative management. Neurourol Urodyn. 2020 Feb;39(2):498-506. doi: 10.1002/nau.24248. Epub 2019 Dec 3. PMID 31794087